CLINICAL TRIAL: NCT07132359
Title: The Mediating Role of Body Image Perception in the Relationship Between Pregnant Women's Attitudes Toward Sexuality and Their Sexual Stress
Brief Title: Role of Body Image in the Relationship Between Pregnant Women's Sexuality and Sexual Stress
Acronym: pregnancy
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ece Kaplan, Asisstant Professor Obstetrics and Gynecology Nursing, University of Gaziantep
Other Study IDs: GAUN-EBE-EKD-04
Record Dates: First submitted 2025-07-25; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Women (Between 18 to 50 Years Old)
Keywords: Body image; attitude toward sexuality; sexual stress; pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Body Understanding Measure for Pregnancy Scale — During the study, the purpose of the study was explained to the pregnant women, and it was stated that participation in the study was completely voluntary and that they could leave the study at any time, and their written and verbal consent was obtained (Informed Consent Form). Pregnant women who agreed to participate in the study filled out the data collection forms individually.

SUMMARY:
Sexual activity is negatively affected during pregnancy. In addition process of adapting to the changes in the pregnant woman's body negatively affects her psychology. Therefore, pregnant woman's perception of her body image can lead to sexual stress. This study aimed to determine the mediating role of body image perception in the relationship between pregnant women's attitudes toward sexuality and their sexual stress. The study sample consisted of 422 pregnant women.

DETAILED DESCRIPTION:
Sexual activity is negatively affected during pregnancy. In addition process of adapting to the changes in the pregnant woman's body negatively affects her psychology. Therefore, pregnant woman's perception of her body image can lead to sexual stress. This study aimed to determine the mediating role of body image perception in the relationship between pregnant women's attitudes toward sexuality and their sexual stress. The study sample consisted of 422 pregnant women. Data collection tools included a "Personal Information Form," the "Attitude Scale toward Sexuality during Pregnancy," the "Female Sexual Distress Scale-Revised" and the "Body Understanding Measure for Pregnancy Scale."

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having no communication problems
* Being at the ≥10th weeks of gestation
* Scoring ≥11.5 on the Female Sexual Distress Scale-Revised

Exclusion Criteria:

* Refusing to participate in the study
* Having been diagnosed with a sexual dysfunction before pregnancy
* Having psychological health problems according to medical records

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study consisted of pregnant women over the age of 20 who presented to the obstetrics and gynecology clinic. During the study, 440 pregnant women were reached. Twelve of them dropped out of the study, and six preferred to have their follow-up at a different hospital; therefore, they were not included in the study. Eventually, the study sample consisted of 422 pregnant women.
Sampling Method: Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
"Attitude Scale toward Sexuality during Pregnancy Scale" | 3 months
  It was conducted with 422 pregnant women. Their written and verbal consent was obtained.
  The Attitude Scale toward Sexuality during Pregnancy: The scale consists of 34 items and three sub-dimensions. The score range of the scale is 34-170. An increase in the scale total score indicates that attitudes toward sexuality during pregnancy are positive.
The Female Sexual Distress Scale-Revised | 3 months
  The scale consists of 13 items to evaluate different aspects of distress related to sexual activity in women. The lowest score that can be obtained from the scale is 0, and the highest is 52. Higher scores indicate higher levels of sexual distress.
The Body Understanding Measure for Pregnancy Scale | 3 months
  The scale consists of 18 items and three sub-dimensions: pregnancy appearance, concerns about weight gain, and physical burden of pregnancy. The score range of the scale is 20-100.As the score increases, the level of dissatisfaction with the perceived body image also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Batuhan Karasin F, Yilmaz T. Psychometric properties of the Turkish version of BUMPs and its relationship with prenatal attachment. J Reprod Infant Psychol. 2025 Jan;43(1):62-75. doi: 10.1080/02646838.2023.2217718. Epub 2023 Jun 5. PMID 37272411